CLINICAL TRIAL: NCT04137822
Title: Expanded Access Program Using IMM-101 for Patients With Advanced Pancreatic Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Impatients N.V. trading as myTomorrows (Industry)
Collaborators: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-IMM101IMM-EU
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Pancreatic Cancer Stage IV; Pancreatic Cancer Stage III
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — IMM-101

INTERVENTIONS:
Biological: IMM-101 — IMM-101 10mg/mL, a suspension of heat-killed whole cell M. obuense in borate-buffered saline. The treatment regimen with IMM-101 is one dose given every 2 weeks for three doses followed by 4 weeks rest, then one dose is given every 2 weeks for a further three doses. Subsequent doses are given every 4 weeks.
  Other Names: Heat-killed whole cell M. obuense

SUMMARY:
An Expanded Access Program for IMM-101 for patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
IMM-101 is a suspension of heat-killed whole cell Mycobacterium obuense. Since it is a heat-killed preparation, treatment is not associated with the potential side-effects of delivering live or attenuated organisms.

Five studies with IMM-101 have been completed including a 110-patient randomised Phase II study in pancreatic cancer and exploratory studies in other solid tumours (melanoma, colorectal cancer and advanced melanoma).

ELIGIBILITY:
Inclusion Criteria:

This Expanded Access Program is available for patients of 18 years or older with advanced pancreatic cancer for whom, in the opinion of their treating physician, other treatment options or clinical trials in this indication are unsuitable.

Exclusion Criteria:

Female patient of child-bearing potential who is not, in the opinion of the physician, using an approved method of birth control (e.g., physical barrier [patient and partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device [IUD]).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- France, Paris, France
- UK, London, United Kingdom

REFERENCES:
- [Background] Costa Neves M, Giakoustidis A, Stamp G, Gaya A, Mudan S. Extended Survival after Complete Pathological Response in Metastatic Pancreatic Ductal Adenocarcinoma Following Induction Chemotherapy, Chemoradiotherapy, and a Novel Immunotherapy Agent, IMM-101. Cureus. 2015 Dec 26;7(12):e435. doi: 10.7759/cureus.435. PMID 26870619
- [Result] Dalgleish AG, Stebbing J, Adamson DJ, Arif SS, Bidoli P, Chang D, Cheeseman S, Diaz-Beveridge R, Fernandez-Martos C, Glynne-Jones R, Granetto C, Massuti B, McAdam K, McDermott R, Martin AJ, Papamichael D, Pazo-Cid R, Vieitez JM, Zaniboni A, Carroll KJ, Wagle S, Gaya A, Mudan SS. Randomised, open-label, phase II study of gemcitabine with and without IMM-101 for advanced pancreatic cancer. Br J Cancer. 2016 Oct 25;115(9):e16. doi: 10.1038/bjc.2016.342. Epub 2016 Oct 11. No abstract available. PMID 27727233